CLINICAL TRIAL: NCT01651429
Title: Multimodal Neuroimaging to Predict Cognitive Resilience Against Sleep Loss
Brief Title: Predicting Cognitive Resilience Against Sleep Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, William Killgore, Assistant Professor, Mclean Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: D12AP00241
Record Dates: First submitted 2012-07-23; First posted 2012-07-27 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Sleep Deprivation
Keywords: Sleep Deprivation
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sleep deprivation (Experimental): Participants will undergo 29 hours of sleep deprivation, 17 of which will be spent in the laboratory.
  Interventions: Behavioral: Sleep deprivation

INTERVENTIONS:
Behavioral: Sleep deprivation — Participants will undergo 29 hours of sleep deprivation. They will wake up at 7:00 am on the day of the study and remain awake in the laboratory until 12:00 pm the next day.

SUMMARY:
Resilience is the ability to cope effectively and adapt to a wide range of stressful environmental challenges. Sleep loss has been shown to reduce activity in the brain regions responsible for resilience. The ability to resist the effects of sleep loss appears to be a stable, trait-like quality. This study will attempt to predict individuals' trait-resistance to sleep loss based on their neurobiology.

DETAILED DESCRIPTION:
Resilience, the ability to cope effectively and adapt to a wide range of stressful environmental challenges, appears to be mediated extensively by the medial prefrontal cortex (MPFC). Sleep deprivation has been shown to reduce metabolic activity throughout the brain, particularly the MPFC. The ability to resist the effects of sleep loss appears to be a stable, trait-like phenomenon that is consistent across situations, suggesting that it may reflect an enduring quality of the underlying neurobiological system. The present study aims to identify the neural basis of resilience and effectively discriminate resistant from vulnerable individuals during an overnight sleep deprivation session. Specifically, the primary aims of this research are 1) to further our understanding of the role of the MPFC in resilience and 2) to develop a statistical prediction algorithm based on multimodal neuroimaging that will reliably discriminate between individuals who are resilient versus vulnerable to the cognitive impairing effects of sleep loss.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-45 years
* Right handedness as assessed by the Edinburgh Handedness Inventory
* For women: regular menstrual cycles (duration between 25 and 35 days with no more than 3 day variation between cycle)

Exclusion Criteria:

* History of head injury with loss of consciousness or post-traumatic amnesia, or major neurological illness
* Medical or neurologic condition that would confound interpretation of results, including alcohol or drug abuse/dependence in the past 6 months, neurological disorders including any history of seizures
* History of cardiac problems
* History of major depressive disorder or anxiety disorder
* Lifetime history of psychotic disorder, including bipolar disorder, schizophrenia, or obsessive compulsive disorder
* Other DSM-IV diagnosis that could affect interpretation of results
* Mixed or left handedness
* Abnormal visual acuity that cannot be corrected by contact lenses
* Daily caffeine use exceeding 400 mg per day
* History of smoking or tobacco use in the past year
* Metal within the body, pregnancy, or other contraindication for MRI procedures
* Use of drugs or medications that could affect functional neuroimaging results (e.g., fluoxetine, beta-blockers)
* Psychotropic medication use within the past 6 weeks

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2013-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Differences in the medial prefrontal cortex (MPFC) as measured by fMRI, DTI, and MRS | Session 2 of study (1 week after enrollment)
  It is hypothesized that, relative to vulnerable individuals, those who are highly resistant to the adverse effects of sleep loss on cognition will show: 1) increased gray matter volume in the MPFC, 2) greater white matter integrity as indicated by the Diffusion Tensor Imaging measure of fractional anisotropy (FA) values in the MPFC, 3) greater functional activation in MPFC during cognitively demanding tasks, 4) greater functional connectivity between MPFC and alerting regions of the midbrain and thalamus; and 5) different ratios of GABA and glutamate within the MPFC.

SECONDARY OUTCOMES:
Psychomotor Vigilance Task (PVT) | At sleep deprivation session (2 weeks after enrollment)
  The PVT will be administered 17 throughout the overnight sleep deprivation session. PVT performance measures participants' alertness and objective resilience to sleep deprivation. PVT performance will be used as a measure to retrospectively assign participants into sleep loss-resistant and sleep loss-vulnerable groups.

OTHER OUTCOMES:
Karolinska Sleepiness Scale (KSS) | At sleep deprivation session (2 weeks after enrollment)
  The KSS will be administered 17 throughout the overnight sleep deprivation session. The KSS provides a measure of subjective sleepiness.

CONTACTS AND LOCATIONS:
Overall Officials: William D Killgore, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States